CLINICAL TRIAL: NCT00532909
Title: A Phase I Trial of Vandetanib Combined With Capecitabine, Oxaliplatin and Bevacizumab for the First-Line Treatment of Metastatic Colorectal Cancer
Brief Title: Phase I Vandetanib Plus Capecitabine, Oxaliplatin and Bevacizumab for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Branimir Sikic (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Branimir Sikic, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COR0006; 97132; COR0006; NCT00532909
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Anal, Colon, and Rectal Cancers; Colorectal Neoplasms; Colon/Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms; Colonic Neoplasms | interventions — vandetanib; Capecitabine; Oxaliplatin; Bevacizumab

INTERVENTIONS:
Drug: Vandetanib — 100mg or 300mg By mouth every day continuous
Drug: Capecitabine — Dosage: 1000mg/m2 By mouth twice a day for 14 days or reduced dose of 800mg/m2 PO BID days1-14.
Drug: Oxaliplatin — dosage: 130mg/m2. IV Day 1 of a 21 day cycle or reduced dose of 100mg/m2 IV Day 1.
Drug: Bevacizumab — Dosage: 7.5mg/kg or 10mg/kg. IV Day 1 (21 day cycle)

SUMMARY:
To determine the maximum tolerated dose of Vandetanib with a current standard first-line chemotherapy regimen, capecitabine and oxaliplatin without and then with bevacizumab for the first line treatment of metastatic colorectal cancer (CRC) and to define the dose limiting toxicities associated with the combination.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent.
* Female and or male age 18 years and over.
* Negative pregnancy test for women of childbearing potential.
* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum.
* Patients with a history of colorectal adenocarcinoma treated by surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease unless an interval of > 5 years has elapsed between the primary surgery and the development of metastatic disease. Clinicians should consider biopsy of lesions to establish diagnosis of metastatic colorectal adenocarcinoma if there is substantial clinical ambiguity regarding the nature or source of apparent metastases.
* A primary or metastatic lesion measurable in at least one dimension by RECIST criteria within 4 weeks prior to entry of study
* WHO performance status of 0-2
* Laboratory values<= 2 weeks prior to randomization:

Absolute Neutrophil Count (ANC) >=1.5 x 10^9/L (>=1500/mm^3) Platelets (PLT) >=100 x 10^9/L (>=100,000/mm^3) Hemoglobin (Hgb) >=9 g/dL Serum creatinine <=1.5 x ULN Serum bilirubin <=1.5 x ULN Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) <=2.5 x ULN (<=5 x ULN if liver metastases present). Note: ERCP or percutaneous stenting may be used to normalize the liver function tests.

Negative or trace for proteinuria based on dip stick reading OR, if documentation of +1 result for protein on dip stick reading, then total urinary protein <=500 mg and measured creatinine clearance (CrCl) >=50 mL/min from a 24-hour urine collection

• Life expectancy >12 weeks

Exclusion Criteria:

• Laboratory results:

Serum bilirubin >1.5 x the upper limit of reference range (ULRR) Serum creatinine >1.5 x ULRR or creatinine clearance >= 50 mL/minute (calculated by Cockcroft-Gault formula.) Potassium <4.0 mmol/L despite supplementation; serum calcium (ionized or adjusted for albumin,) or magnesium out of normal range despite supplementation.

Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x ULRR or alkaline phosphatase (ALP) >2.5 x ULRR, or >5x ULRR if judged by the investigator to be related to liver metastases

* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
* Clinically significant cardiac event such as myocardial infarction; New York Heart Association (NYHA) classification of heart disease >= 2 within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
* History of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication, is not excluded.
* Previous history of QTc prolongation as a result from other medication that required discontinuation of that medication.
* Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age.
* Presence of left bundle branch block (LBBB.)
* QTc with Bazett's correction that is unmeasurable, or <480 msec on screening ECG. If a patient has QTc >= 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be <480 msec in order for the patient to be eligible for the study.)
* Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce CYP3A4 function
* Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
* Currently active diarrhea that may affect the ability of the patient to absorb the vandetanib or tolerate diarrhea.
* Women who are currently pregnant or breastfeeding.
* Previous or current malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Receipt of any investigational agents within 30 days prior to commencing study treatment
* Last dose of prior chemotherapy discontinued less than 4 weeks before the start of study therapy
* Last radiation therapy within the last 4 weeks before the start of study therapy, except palliative radiotherapy
* Any unresolved toxicity greater than CTC grade 1 from previous anti-cancer therapy
* Previous enrollment or randomization of treatment in the present study
* Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of vandetanib in combination with capecitabine, oxaliplatin and bevacizumab | Following treatment

SECONDARY OUTCOMES:
Effect of vandetanib on the pharmacokinetics (PK) of capecitabine and oxaliplatin | During and following treatment
Effects of this treatment on tumor remission, progression free survival, and overall survival of patients | Following treatment
Dose limiting toxicities associated with the combination | During and following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Branimir I Sikic, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States